CLINICAL TRIAL: NCT03612219
Title: A Multicenter, Phase II Clinical Study of Adjuvant Apatinib After IMRT With Concurrent Chemotherapy Versus IMRT With Concurrent Chemotherapy in High-risk Metastasis of Nasopharyngeal Carcinoma
Brief Title: Adjuvant Treatment of Apatinib in Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Jiang (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); Guangxi Minzu Hospital (Unknown); People's Hospital of Lingshan (Unknown); Guangxi Naxishan Hospital (Other); People's Hospital of Baise (Unknown); Laibin People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Wei Jiang, Wei Jiang, MD, PhD, Guilin Medical University, China
Organization: Guilin Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLMU-04
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Apatinib; Adjuvant treatment; Progression-free survival
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — apatinib; Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMRT with CC+Adjuvant Apatinib (Experimental): Treat with Apatinib mesylate tablet for adjuvant treatment(the dose was 250 mg,orally,qd,28 days for an observation period,Six cycles)of local advanced nasopharyngeal carcinoma after Intensity-modulated radiation therapy (IMRT) with concurrent chemotherapy(cisplatin).
  Interventions: Drug: Apatinib mesylate tablet; Radiation: Intensity-modulated radiation therapy (IMRT); Drug: Cisplatin
- IMRT with CC (Active Comparator): Only obeservation after Intensity-modulated radiation therapy (IMRT) with concurrent chemotherapy(cisplatin).
  Interventions: Radiation: Intensity-modulated radiation therapy (IMRT); Drug: Cisplatin

INTERVENTIONS:
Drug: Apatinib mesylate tablet — Adjuvant treatment by apatinib mesylate tablet to local advanced nasopharyngeal carcinoma after IMRT with concurrent chemotherapy.the dose of apatinib mesylate tablet was 250 mg,orally,qd,28 days for an observation period,six cycles.
  Other Names: No.
  Arms: IMRT with CC+Adjuvant Apatinib
Radiation: Intensity-modulated radiation therapy (IMRT) — Intensity-modulated radiation therapy (IMRT):GTVnx 69.69Gy, GTVnd 60-68Gy, PTV1 59.4Gy and PTV2 54Gy in 33 fractions, 5 days/week.
  Other Names: No.
Drug: Cisplatin — Concurrent chemotherapy: patients received intravenous cisplatin 80mg/m2(D1-3), 3-week chemotherapy for 3 cycles.
  Other Names: No.

SUMMARY:
The study is to evaluate the efficacy and safety of apatinib for adjuvant treatment of High-risk metastasis of nasopharyngeal carcinoma after IMRT with concurrent chemotherapy,including progression-free survival (PFS),evaluation of drug safety.,and overall survival (OS),distant metastasisfree survival (DMFS),locoregional relapse-free survival (LRRFS),and quality of life score (QoL).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Ⅰ.To determine if adjuvant apatinib after IMRT with concurrent chemotherapy is better to only obeservation after IMRT with concurrent chemotherapy for progression-free survival in High-risk metastasis of nasopharyngeal carcinoma.

SECONDARY OBJECTIVES:

Ⅰ.To explore the adjuvant medication regimen of local advanced nasopharyngeal carcinoma after IMRT with concurrent chemotherapy.

Ⅱ.Provide high-level evidence-based medical evidence for the new individualized treatment strategy of nasopharyngeal carcinoma patients.

OUTLINE:

Patients are randomized to one of the two treatment arms.

ARM 1: treat with apatinib(the dose was 250 mg,orally,qd,28 days for an observation period,Six cycles) for adjuvant treatment of local advanced nasopharyngeal carcinoma after IMRT with concurrent chemotherapy.

ARM 2:only obeservation after IMRT with concurrent chemotherapy. IMRT: GTVnx 69.69Gy, GTVnd 60-68Gy, PTV1 59.4Gy and PTV2 54Gy in 33 fractions, 5 days/week.

Concurrent chemotherapy:Cisplatin 80mg/m2(D1-3), 3-week chemotherapy for 3 cycles.

After completion of study therapy, patients are followed up every 3-4 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type) Tumor staged as T4 or N2-3 or lymph node>3cm and M0(according to the 8th AJCC edition).
2. Adequate hematological function: hemoglobin >80 g/L, neutrophil count > 1.5×10^9/L, platelet count 80×10^9/L.
3. Adequate liver function (serum transminase ≤ 2.5 times higher than upper limit),adequate renal function (creatinine clearance ≥ 60 mL/min).
4. Karnofsky performance status (KPS) score of at least 70 or Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Patients must give signed informed consent.

Exclusion Criteria:

1. Other or mixed pathological type.
2. age > 70 years.
3. Severe heart, liver and kidney damage.
4. History of other malignancy.
5. Prior chemotherapy or radiation of the primary tumor.
6. History of psychiatric disorders.
7. Positive urine protein.
8. A healed wound for long time or incomplete fracture.
9. Before treatment,MRI showed that the tumor might be an important risk factor (for example, wrapping around the internal carotid artery / vein); or researchers judged that the tumor is a high risk of serious blood vessel bleeding during the treatment.
10. Patient who has high blood pressure can not be controlled by a single antihypertensive drug treatment (Systolic pressure > 140 mmHg, diastolic pressure > 90 mmHg.
11. Any unstable angina pectoris;with a history of angina pectoris were newly diagnosed with angina pectoris within 3 months before screening; any myocardial infarction events occurred within 6 months before screening; arrhythmia (including QTcF: male ≥ 450ms, female ≥ 470 ms) need long time use of antiarrhythmic drugs and heart function insufficiency ≥II according to New York Heart Association class.
12. Medical history of arteriovenous thrombosis event within the past year, such as cerebral vascular accident (including transient ischemic attack) and deep venous thrombosis (venous catheter thrombosis caused by chemotherapy and investigator judged that the patient had recovered, these patients should be except) and pulmonary embolism.
13. Patient who has serious hemorrhages, any serious bleeding events classification at 3 degree or more (according to CTCAE4.0) within the last 4 weeks.
14. Patient who has abnormal coagulation and bleeding tendency (signed informed consent before 14 days, and must be satisfied: INR is in the normal range without the use of anticoagulants); Application of anticoagulants or vitamin K antagonists such as Hua Falin, heparin or its analogues, with international normalized ratio (INR) is less than 1.5, allows the use of small dose Hua Falin (1 mg orally, once daily) or small dose aspirin (total dose ≤ 100 mg daily).
15. For females:patients should be surgical sterilization or postmenopausal patients, or willing to receive a medical approved contraception during treatment and 6 months after the end of the treatment; serum or urine pregnancy test must be negative, and must be non lactating period within 7 days before study; for males: patients should be treated with surgical sterilization or willing to receive a medical approved contraception during treatment and 6 months after the end of the treatment.
16. Any factors that affect the oral drug, such as the inability to swallow, diarrhea and intestinal obstruction.
17. Medical history of immunodeficiency, or other acquired, congenital immunodeficiency disease, or history of organ transplantation.
18. Any serious harm to the subject's safety or evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-07-28 (Estimated); Study Completion 2021-07-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  The time from the first day of therapy to locoregional relapse, distant relapse or tumor-related death

SECONDARY OUTCOMES:
Overall survival | 3 years
  The time from the first day of therapy to death or last follow-up
Locoregional relapse-free survival | 3 years
  The time from the first day of treatment to the time of first locoregional relapse
Distant metastasis-free survival | 3 years
  The time from the first day of treatment to the time of first distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, Ph.D., Study Director — Guilin Medical University, China
Locations (6):
- China (6):
  - People's Hospital of Baise, Baise City, Guangxi
  - Guangxi Naxishan Hospital, Guilin, Guangxi
  - Guilin Medical University, Guilin, Guangxi
  - People's Hospital of Laibin, Laibin, Guangxi
  - People's Hospital of Lingshan, Linshan, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi